CLINICAL TRIAL: NCT05378581
Title: Evaluation of the Use of a Virtual Reality Mask During Blood Tests and Prick Tests Performed in Allergic Children Aged 7 to 13 Years: a Multicenter, Randomized Trial
Brief Title: Use of Virtual Reality Mask During Blood and Skin Allergic Tests in 7 to 13 Children
Acronym: REVAPRICK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GIRCI 2020 USCLADE; 2021-A02125-36 (Other: ANSM)
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Children, Only; Pain, Procedural; Anxiety and Fear
Keywords: virtual reality mask; children from 7 to 13; allergic pricks tests; consultation and pediatric's day hospital
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, two arms parallel, multicenter therapeutic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard (Active Comparator): Use local anesthesic cream + nurse or parents distraction +/- anesthesic or anxiolytic gas
  Interventions: Other: control arm
- virtual reality (Experimental): Use local anesthesic cream and virtual reality mask
  Interventions: Device: Virtual reality mask

INTERVENTIONS:
Device: Virtual reality mask — virtual reality mask Deepsen® with age-appropriate software Birdy®
  Arms: virtual reality
Other: control arm — usual process
  Arms: standard

SUMMARY:
Main objective :

Evaluate the effect of using a virtual reality mask during the blood test and pricks tests in allergic children aged from 7 to 13 years.

Hypothesis :

Using virtual reality mask during blood test and pricks tests for allergic kids from 7 to 13 would reduce anxiety and pain

DETAILED DESCRIPTION:
Investigation of food or respiratory allergy is based on prick tests and serum specific immunoglobulin E assays. The nurse often controls the blood test pain but during the skin tests, many children cry, feeling both fear and pain. This traumatic experience will in most cases be repeated during the child's allergic follow-up.

To date, there are few effective means of limiting anxiety and pain associated with prick tests and therefore little research work on this subject.

Immersion in virtual reality (VR) seems to be an interesting way of distraction for children from 7 to 13 years needing this treatment. Indeed, it makes it possible to saturate the sensorially of the child thus reducing the nociceptive perceptions and the anxiety. The choice of VR mask with pediatric program specific seems interesting for this children This is a randomized, open-label, two-armed parallel, multicenter therapeutic trial comparing an analgesic strategy using authorized medical devices (conventional strategy) with a virtual reality mask distraction technique for allergics tests in children from 7 to 13 years old hospitalized in the pediatric consultation of Clermont Ferrand University Hospital and in the day hospital of Saint-Etienne University Hospital

The control arm is the local anesthetic cream (for the blood test) arm with distraction from nurse/parents +/-anesthesic and anxiolytic gas and the experimental arm is the local anesthetic cream + virtual reality mask distraction

The nurse informs and obtains the consent of the child and his parents. Then she measures child's pain and anxiety before the care, during the blood test, at the third prick test and immediately after the care.

She also notes the anxiety of the parents before and after the care. Finally, the satisfaction of the child, parents, nurses will be collected at the end of the care.

After statistical analysis of these two arms, it will be possible to determine the value of the virtual reality mask to reduce the child's pain and anxiety during the pricks tests.

ELIGIBILITY:
Inclusion Criteria:

* Children from 7 to 13 years old requiring blood test and prick tests in pediatric consultation at the Clermont-Ferrand University Hospital and in the pediatric's day hospital at the Saint-Etienne University Hospital
* Subjects and their parents who were informed about the study and gave informed consent
* Enrollment in the Social Security system
* Children and parents able to use the self-report scales proposed in the study

Exclusion Criteria:

Children from 7 to 13 :

* presenting a contraindication to the use of the virtual reality mask: heart disease, epilepsy, psychiatric illness (major anxiety, post-traumatic stress disorder)
* Having a modification of pain's integration (spina bifida for example)
* Having received an analgesic before the care
* Requiring contact isolation
* With a history of seizures or motion sickness
* Refusal of the parents and/or the child

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
children's pain hetero-evaluation | during blood test
  children's pain evaluation by the nurse with the visual analog scale quote from 0 to 10, 10=worst score
children's pain hetero-evaluation | during procedure (prick test)
  children's pain evaluation by the nurse with the visual analog scale from 0 to 10, 10= worst score
children's pain self-evaluation | 5 min after the care
  self evaluation of children's pain with the visial analog scale in vertical position quote from 0 to 10, 10=worst score

SECONDARY OUTCOMES:
change from baseline children's anxiety at just after the care | before the care and 5 min after the care
  self-evaluation of children's anxiety with the scale "child fear scale" quote from 0 to 4, 4= worst score
children's anxiety hetero evaluation | during blood test
  children's anxiety evaluation by the nurse with the scale "child fear scale" quote from 0 to 4, 4= worst score
children's anxiety hetero evaluation | during procedure (prick tests)
  children's anxiety evaluation by the nurse with the scale "child fear scale" quote from 0 to 4, 4= worst score
change from baseline parents' anxiety at just after the care | before the care and 5 min after the care
  self-evaluation of parents' anxiety with the numerical scale quote from 1 to 10, 10= worst score
evaluation of the care | 5 min after the care
  satisfaction of the care for children, parents and nurses with satisfaction questionnaire for children : a score from 1 to 3 (3=best score, very satisfied) for parents with a score from 1 to 5 (5= best score, very satisfied) and for nurse with a score from 1 to 5 (5= best score, very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra USCLADE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No